CLINICAL TRIAL: NCT04048252
Title: Development of a Therapeutic Education Program for Patients With Metastatic Prostate Cancer Treated With New Generation Hormone Therapy: Construction and Feasibility Study
Brief Title: Development of a Therapeutic Education Program for Patients With Metastatic Prostate Cancer Treated With New Generation Hormone Therapy
Acronym: PROSTED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2019/NH-02
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Focus group
  Interventions: Other: Focus group creation
- Workshop
  Interventions: Other: Workshop

INTERVENTIONS:
Other: Focus group creation — Patients will join with researchers for a 2 hour recorded group discussion to highlight themes identified to require educational intervention
  Groups: Focus group
Other: Workshop — Patients will attend 3-4 workshops on eg disease knowledge, medication management and side effects, adapted physical activity and nutrition
  Groups: Workshop

SUMMARY:
The development of a personalized therapeutic education program dedicated to patients with metastatic prostate cancer and receiving next-generation hormone therapy would improve their knowledge of the disease, medication adherence and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic prostate cancer treated with enzalutamide or abiraterone acetate for at least 3 months
* The patient must have given their free and informed consent and signed the consent form
* The patient must be insured or the beneficiary of an insurance policy

Exclusion Criteria:

* The subject is not in a fit state to express their consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic prostate cancer and receiving next-generation hormone therapy
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Create a focus group | Day 0
  Transcribe interview and mark key points
Patient satisfaction | End of workshops (max 2 months)
  Yes/no
Successful running of workshop | End of workshops (max 2 months)
  Yes/no evaluated by the workshop leader

SECONDARY OUTCOMES:
Patient participation rate in workshops | End of workshops (max 2 months)
Patient-reported acceptability of programme | End of workshops (max 2 months)
  In-house questionnaire: 4 questions on 0-5 scale unacceptable to very acceptable and 4 open questions
Patient-reported satisfaction of programme | End of workshops (max 2 months)
  In-house questionnaire: 5 questions on 0-5 scale unsatisfied to very satisfied
Patient knowledge of their disease | End of workshops (max 2 months)
  In-house quiz: 7 multiple-choice questions
Patient quality of life | 1 month after last workshop
  EQ-5D-3L
Patient medication adherence | End of workshops (max 2 months)
  MMAS-9 questionnaire: good adherence is score = 8

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Houede, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France